CLINICAL TRIAL: NCT05484297
Title: Increasing Social Connection Through Crisis Caring Contacts: A Pragmatic Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDR 21-087; 1I01HX003428-01 (NIH)
Record Dates: First submitted 2022-07-12; First posted 2022-08-02 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Loneliness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either the intervention or the control group. Block-randomization schemes using random block sizes to assign the two study arms will be created in R using the blockrand package before study start. Randomization will be stratified by study site. The intervention will consist of a series of post cards with Crisis Caring Contacts content sent over 10 months. The control group will receive similar post cards intended to control for attention received but not including elements thought to be "active ingredients" in the intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Following recommendations for blinding in behavioral interventions, participants will be blinded by limiting details about the study hypotheses and differences between the study arms. Furthermore, research staff involved in outcome assessment and study biostatisticians involved in data analysis will be blinded to study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment arm will receive the intervention post cards
  Interventions: Behavioral: Crisis Caring Contacts post cards
- Control (Sham Comparator): Participants in the control arm will receive the control post cards
  Interventions: Behavioral: Control post cards

INTERVENTIONS:
Behavioral: Crisis Caring Contacts post cards — A series of post cards with Crisis Caring Contacts content sent over 10 months
  Arms: Treatment
Behavioral: Control post cards — A series of post cards intended to control for attention received but not including elements thought to be "active ingredients" in the intervention
  Arms: Control

SUMMARY:
The main purpose is to learn if sending messages from the VA (called "Caring Contacts") reduces loneliness and improves mental health. The investigators want to understand if these messages are effective in Veterans aged 60 and above who have missed appointments at the VA even though they have health problems. Participants will receive up to 10 postcards mailed in envelopes from a fellow Veteran (Peer Specialist) from their local VA, and will be asked to fill out four surveys. The investigators are recruiting 920 Veterans aged 50 years and older who have felt isolated and have missed appointments at the VA to join this study.

DETAILED DESCRIPTION:
Lack of social connection is a common and powerful predictor of suicidal ideation, suicide attempts, functional decline, and death, even after adjustment for sociodemographic and clinical variables. Loneliness, specifically, is associated with a 26% increased likelihood of all-cause mortality. The urgency of addressing these problems is only amplified by the COVID-19 pandemic, which for some time may further increase loneliness, suicide, and other causes of mortality. Due to their risk for loneliness and negative health outcomes, a group of particular concern is older adults and patients with medical or psychiatric comorbidity who have poor treatment engagement.

Caring Contacts is an intervention that can address loneliness and treatment disengagement. It involves periodically sending brief messages to at-risk individuals with nondemanding expressions of care and concern. It is one of just two non-pharmacologic interventions to have evidence in randomized controlled trials (RCTs) for reducing rates of suicide. However, Caring Contacts has only been evaluated in a relatively narrowly indicated population of patients with acute psychiatric issues.

Major gaps in the understanding of Caring Contacts include whether it reduces loneliness, whether it can diminish causes of mortality besides suicide, and whether it is effective older Veterans and patients with treatment disengagement. The overarching objective of this project is to evaluate "Crisis Caring Contacts" (CCC), an adaptation of Caring Contacts tailored to Veterans at risk for lack of social connection and lapses in treatment amidst the COVID-19 pandemic and its aftermath.

Primary aims for this study are: 1) Among older Veterans with poor treatment engagement, evaluate the effectiveness of Crisis Caring Contacts in decreasing loneliness, compared to enhanced usual care; 2) Evaluate the effect of Crisis Caring Contacts on other important outcomes, including treatment engagement and suicidal ideation; 3) Explore potential moderators of treatment response to Crisis Caring Contacts; and 4) Explore the effect of Crisis Caring Contacts on all-cause mortality, suicide attempts, and drug overdoses.

Impact: This project will advance scientific understanding of key gaps related to the mechanisms and outcomes of Caring Contacts, while also evaluating a timely, pragmatic, low-cost, and scalable intervention for Veterans affected by lack of social connection and treatment engagement.

ELIGIBILITY:
Inclusion Criteria:

* age 50 years and above
* have at least four VA appointments in the prior 6-18 months in primary care or mental health
* have at least two comorbidities contained in the Elixhauser Index
* a) zero completed appointments in the past 6 months and zero appointments scheduled, or b) in the 90th percentile or higher in terms of no-shows or appointments canceled by patient in the prior 12 months

Exclusion Criteria:

* no valid mailing address
* no valid phone number
* inclusion in an existing Caring Contacts program
* diagnosis of neurocognitive disorder or other significant cognitive impairment indicative of inadequate decision-making capacity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
UCLA Loneliness Scale, Version 3 | 12-month follow-up
  This scale has a score range from 20 -80, with higher scores representing greater degrees of loneliness.
Count of mental health or primary care visits over 12 months | The 12-month period from the date of randomization to 12-month follow-up
  Treatment engagement will be assessed by counting VA outpatient visits to mental health or primary care during the 12 months after randomization. More visits will represent greater treatment engagement.

SECONDARY OUTCOMES:
PROMIS Short Form v2.0 - Emotional Support 4a | 12-month follow-up
  This scale has a range from 4 - 20, with higher scores representing greater perceived emotional support.
Trust in Public Healthcare System, Institutional Trust Subscale (adapted for VA) | 12-month follow-up
  Adapted to assess trust in the VA specifically, this scale has a score range from 3 - 15, with higher scores representing more trust.
Depressive Symptom Index Suicidality Subscale (DSI-SS) | 12-month follow-up
  This scale has a score range from 0 - 12, with higher scores representing greater degrees of suicidality.
Suicide Ideation Scale (SIS) | 12-month follow-up
  This scale has a score range from 10 - 50, with higher scores representing greater degrees of suicidality.

CONTACTS AND LOCATIONS:
Overall Officials: Alan R. Teo, MD MS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (3):
- United States (3):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Das A, Padala KP, Crawford CG, Teo A, Mendez DM, Phillips OA, Wright BC, House S, Padala PR. A systematic review of loneliness and social isolation scales used in epidemics and pandemics. Psychiatry Res. 2021 Dec;306:114217. doi: 10.1016/j.psychres.2021.114217. Epub 2021 Oct 8. PMID 34644661
- [Result] Hynes DM, Niederhausen M, Chen JI, Shahoumian TA, Rowneki M, Hickok A, Shepherd-Banigan M, Hawkins EJ, Naylor J, Teo A, Govier DJ, Berry K, McCready H, Osborne TF, Wong E, Hebert PL, Smith VA, Bowling CB, Boyko EJ, Ioannou GN, Iwashyna TJ, Maciejewski ML, O'Hare AM, Viglianti EM, Bohnert AS. Risk of Suicide-Related Outcomes After SARS-COV-2 Infection: Results from a Nationwide Observational Matched Cohort of US Veterans. J Gen Intern Med. 2024 Mar;39(4):626-635. doi: 10.1007/s11606-023-08440-9. Epub 2023 Oct 26. PMID 37884839

DOCUMENTS (1):
  • Informed Consent Form (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT05484297/ICF_000.pdf